CLINICAL TRIAL: NCT05208775
Title: A Phase III, Randomized, Controlled Study of Endoscopic Submucosal Dissection Versus Photodynamic Therapy for Early Esophageal Cancer
Brief Title: A Comparative Study of Endoscopic Submucosal Dissection and Photodynamic Therapy for Early Esophageal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Henan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ECPDT-002
Record Dates: First submitted 2022-01-10; First posted 2022-01-26 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2021-12

CONDITIONS: Esophageal Carcinoma in Situ AJCC V7
Keywords: Early esophageal carcinoma; Photodynamics Therapy; Endoscopic submucosal dissection
MeSH Terms: conditions — Esophageal Neoplasms | interventions — 1-phenyl-3,3-dimethyltriazene; Endoscopic Mucosal Resection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PDT group (Experimental): After enrollment, patients were injected with photosensitizer at a dose of 2mg/kg, and received photodynamic irradiation 48 hours later.
  Interventions: Procedure: PDT
- ESD group (Active Comparator): Patients received standard ESD treatment after enrollment
  Interventions: Procedure: ESD

INTERVENTIONS:
Procedure: PDT — Drug: (Hematoporphyrin sodium injection) Hematoporphyrin sodium injection (xibofen):2mg/kg I.V.
  Laser irradiation:
  48 hours after the patient input the photosensitizer, the laser irradiation time is 900 seconds, and the output power is 200 watts.
  Other Names: Photodynamics Therapy
  Arms: PDT group
Procedure: ESD — The patients received standard endoscopic submucosal dissection after enrollment.
  Other Names: Endoscopic submucosal dissection
  Arms: ESD group

SUMMARY:
The purpose of this study was to compare the efficacy and safety of Photodynamic therapy (PDT) and Endoscopic submucosal (ESD) dissection in the treatment of early esophageal cancer.

DETAILED DESCRIPTION:
Background: Photodynamic therapy (PDT) is recommended by the NCCN guidelines as an effective method for the treatment of early esophageal cancer. However, there is no clinical trial data so far on whether its efficacy can be compared with that of standard Endoscopic submucosal (ESD). Our team will conduct a detailed study on it.

Aim: to compare the efficacy and safety of Photodynamic therapy (PDT) and Endoscopic submucosal (ESD) dissection in the treatment of early esophageal cancer.

Methods: This study intends to recruit 46 patients with early esophageal cancer and randomly divide them into two groups: one group to receive ESD and the other group to receive PDT.The efficacy and safety were observed after 2 years of follow-up.

Primary endpoints: The recurrence rates at 3 months, 6 months, and 2 years were compared.

ELIGIBILITY:
Inclusion Criteria:

* High-grade intraepithelial neoplasia of the esophagus
* 18-80 years old
* The tumor was confined to the lamina propria of the mucosa
* The tumor invaded the submucosa and was limited to 200 microns

Exclusion Criteria:

* The tumor invaded the entire circumference of the esophagus
* The tumor invaded the muscularis or submucosa more than 200 microns
* The patient has difficulty tolerating anesthesia due to other diseases
* Pregnant or breastfeeding women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
2-year disease-free survival rate | 2 year
  The percent of 2 year disease-free survival after random allocation, percent

SECONDARY OUTCOMES:
Esophageal stenosis rate at 3 months | 3 months
  Stenosis rate of esophagus after 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Shegan Gao, MD, PhD, Study Chair — The First Affiliated Hospital and College of Henan University of Science and Technology; Tanyou Shan, MD, PhD, Study Director — The First Affiliated Hospital and College of Henan University of Science and Technology; Lijuan Wu, MD, PhD, Study Director — The First Affiliated Hospital and College of Henan University of Science and Technology; Caihong Dong, MD，PhD, Principal Investigator — The First Affiliated Hospital and College of Henan University of Science and Technology; Jiachun Sun, MD, PhD, Principal Investigator — The First Affiliated Hospital and College of Henan University of Science and Technology; Wanying Li, MD, Principal Investigator — The First Affiliated Hospital and College of Henan University of Science and Technology; Xiaozhi Yuan, MD, PhD, Principal Investigator — The First Affiliated Hospital and College of Henan University of Science and Technology; Mengxi Zhang, MD, Principal Investigator — The First Affiliated Hospital and College of Henan University of Science and Technology

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yano T, Minamide T, Takashima K, Nakajo K, Kadota T, Yoda Y. Clinical Practice of Photodynamic Therapy Using Talaporfin Sodium for Esophageal Cancer. J Clin Med. 2021 Jun 24;10(13):2785. doi: 10.3390/jcm10132785. PMID 34202917
- [Background] National Health Commission Of The People's Republic Of China. Chinese guidelines for diagnosis and treatment of esophageal carcinoma 2018 (English version). Chin J Cancer Res. 2019 Apr;31(2):223-258. doi: 10.21147/j.issn.1000-9604.2019.02.01. No abstract available. PMID 31156297
- [Background] Zeng R, Liu C, Li L, Cai X, Chen R, Li Z. Clinical Efficacy of HiPorfin Photodynamic Therapy for Advanced Obstructive Esophageal Cancer. Technol Cancer Res Treat. 2020 Jan-Dec;19:1533033820930335. doi: 10.1177/1533033820930335. PMID 32578508
- [Background] Yoon HY, Cheon YK, Choi HJ, Shim CS. Role of photodynamic therapy in the palliation of obstructing esophageal cancer. Korean J Intern Med. 2012 Sep;27(3):278-84. doi: 10.3904/kjim.2012.27.3.278. Epub 2012 Sep 1. PMID 23019392
- [Background] Itabashi M, Nasierowska-Guttmejer A, Shimoda T, Majewski P, Rezner W, Sikora K, Srutek E, Steplewska K, Swatek J, Szumilo J, Wierzchniewska-Lawska A, Wronecki L, Zembala-Nozynska E, Arai T, Fujita M, Kawachi H, Unakami M, Kamoshida T. The importance of the concept and histological criteria of "intraepithelial squamous cell carcinoma" of the esophagus: in comparison between Western and Japanese criteria. Esophagus. 2017;14(4):333-342. doi: 10.1007/s10388-017-0583-7. Epub 2017 Jun 14. PMID 28983230
- [Background] Zheng JY, Chen YH, Chen YY, Zheng XL, Zhong SS, Deng WY, Zheng JH, Guo XB, Gao LY, Liang W. Presence of pink-color sign within 1 min after iodine staining has high diagnostic accordance rate for esophageal high-grade intraepithelial neoplasia/invasive cancer. Saudi J Gastroenterol. 2019 Mar-Apr;25(2):113-118. doi: 10.4103/sjg.SJG_274_18. PMID 30588952
- [Background] Omae M, Hagstrom H, Ndegwa N, Vieth M, Wang N, Vujasinovic M, Baldaque-Silva F. Wide-field endoscopic submucosal dissection for the treatment of Barrett's esophagus neoplasia. Endosc Int Open. 2021 May;9(5):E727-E734. doi: 10.1055/a-1386-3668. Epub 2021 Apr 22. PMID 33937514
- [Background] Wu W, Wu YL, Zhu YB, Wei Q, Guo Y, Zhu ZG, Yuan YZ. Endoscopic features predictive of gastric cancer in superficial lesions with biopsy-proven high grade intraepithelial neoplasia. World J Gastroenterol. 2009 Jan 28;15(4):489-95. doi: 10.3748/wjg.15.489. PMID 19152456
- [Background] Ke Y, van Munster SN, Xue L, He S, Zhang Y, Dou L, Liu Y, Liu X, Liu Y, Li W, Lv N, Dawsey SM, Weusten BLAM, Bergman JJGHM, Wang G. Prospective study of endoscopic focal cryoballoon ablation for esophageal squamous cell neoplasia in China. Gastrointest Endosc. 2019 Aug;90(2):204-212. doi: 10.1016/j.gie.2019.03.017. Epub 2019 Mar 25. PMID 30922862